CLINICAL TRIAL: NCT00422734
Title: Tadalafil 5 mg Once a Day Compared to Placebo in Improving Erectile Dysfunction and Sexual Quality of Life
Brief Title: Tadalafil Taken Daily Compared to Placebo on Improvement of Getting and Maintaining an Erection and Sexual Quality of Life
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9501; H6D-MC-LVGH
Record Dates: First submitted 2007-01-16; First posted 2007-01-17 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Active Comparator): 5 mg tadalafil
  Interventions: Drug: tadalafil

INTERVENTIONS:
Drug: tadalafil — 5 mg tadalafil tablet taken by mouth once a day for 12 weeks
  Other Names: LY450190; Cialis; IC351
  Arms: 2
Drug: Placebo — placebo tablet taken by mouth once a day for 12 weeks
  Arms: 1

SUMMARY:
To determine if tadalafil 5 mg daily compared to placebo when given for 12 weeks improves getting and maintaining an erection in men with erectile dysfunction and if there are improvements in the sexual quality of life of the man and his female study partner

ELIGIBILITY:
Inclusion Criteria:

Male

* History of erectile dysfunction (ED) for at least 3 months duration
* Anticipate having the same female partner willing to participate throughout the study
* At least 18 years of age at Visit 1 and agree to make at least 4 sexual attempts during the early phase of the study
* Adequate partner sexual function as determined by a Female Sexual Function Index
* Willing to record responses to efficacy questionnaires, sexual quality of life questionnaires and other instruments used in the study

Exclusion Criteria:

* May not participate in the study if you have taken tadalafil previously.
* History of cardiac conditions including angina requiring treatment with nitrates, heart disease of coronary conditions including myocardial infarction, bypass surgery, angioplasty or stent placement for specified time before starting the study.
* Have sexual partner not willing to complete the scales.
* Use of nitrates.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (19):
- United States (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntsville, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newport Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stuart, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Virginia Beach, Virginia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salzburg, Austria
- France (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augsburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leverkusen
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Joya, Mexico

REFERENCES:
- [Derived] Porst H, Gacci M, Buttner H, Henneges C, Boess F. Tadalafil once daily in men with erectile dysfunction: an integrated analysis of data obtained from 1913 patients from six randomized, double-blind, placebo-controlled, clinical studies. Eur Urol. 2014 Feb;65(2):455-64. doi: 10.1016/j.eururo.2013.09.037. Epub 2013 Oct 2. PMID 24119319
- [Derived] Shabsigh R, Seftel AD, Kim ED, Ni X, Burns PR. Efficacy and safety of once-daily tadalafil in men with erectile dysfunction who reported no successful intercourse attempts at baseline. J Sex Med. 2013 Mar;10(3):844-56. doi: 10.1111/j.1743-6109.2012.02898.x. Epub 2012 Oct 4. PMID 23035781
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Tadalafil
Started | 78 | 264
Completed | 64 | 243
Not Completed | 14 | 21
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 1 | 6
Not completed — Withdrawal by Subject | 12 | 8
Not completed — Adverse Event | 0 | 3
Not completed — Partner Decision | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tadalafil | Total
Number analyzed (Participants) | 78 | 264 | 342
Age Continuous [Mean (Standard Deviation); unit: years] | 53.82 (10.72) | 54.42 (10.04) | 54.29 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 78 | 264 | 342
Region of Enrollment [Number; unit: participants]
  France | 11 | 41 | 52
  United States | 29 | 107 | 136
  Mexico | 19 | 63 | 82
  Austria | 8 | 17 | 25
  Germany | 11 | 36 | 47
Erectile Dysfunction History - Duration [Number; unit: participants]
  >= 1 year | 73 | 240 | 313
  >= 3 months and < 6 months | 1 | 8 | 9
  >= 6 months and < 1 year | 4 | 16 | 20
Erectile Dysfunction History - Etiology [Number; unit: participants]
  Mixed | 34 | 114 | 148
  Organic | 29 | 91 | 120
  Psychogenic | 12 | 30 | 42
  Unknown | 3 | 29 | 32
International Index of Erectile Function (IIEF) - Erectile Dysfunction Severity [Number; unit: participants]
  Mild (17-30) | 35 | 123 | 158.0
  Moderate (11-16) | 22 | 71 | 93.0
  Severe (1-10) | 20 | 63 | 83.0
  Missing | 1 | 7 | 8.0
Race/Ethnicity [Number; unit: participants]
  African | 0 | 6 | 6
  Caucasian | 57 | 188 | 245
  Hispanic | 21 | 69 | 90
  Native American | 0 | 1 | 1
International Index of Erectile Function (IIEF) - Erectile Function Domain [Mean (Standard Deviation); unit: units on a scale] — Self-reported erectile function over the past 4 weeks. Scores range from 0 (low or no erectile function) to 5 (high erectile function) on 6 questions (1-5, 15 of the IIEF). Total Erectile Function Domain scores range from 0 to 30.
  units on a scale | 15.27 (6.49) | 15.73 (6.13) | 15.62 (6.21)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Endpoint in the International Index of Erectile Function (IIEF)- Erectile Function Domain Score (Sum of IIEF Questions 1-5 and 15)
Description: Measures erectile function over the past 4 weeks on Questions 1-5 and 15 (6 questions) of the International Index of Erecile Function (IIEF) questionnaire. Scores range from 0 (low/no erectile function) to 5 (high erectile function), thus the 6 questions of the IIEF-EF domain range from 0 to 30.
Time Frame: Baseline and 12 weeks
Population: last observation carried forward for all randomized participants having both baseline and at least one post-baseline data measurement
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 72 | 244
units on a scale | 0.49 (0.781) | 8.03 (0.449)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; The null hypotheses (no treatment effect with respect to IIEF EF domain or SEP2 or SEP3) were each tested at a specified level of 0.05. In order to pass a serial gatekeeper, it was necessary to reject all three hypotheses. The two null hypotheses (no treatment effect with respect to subject SLQQ-SQoL domain and no treatment effect with respect to partner SLQQ-SQoL domain) were then each tested at a significance level of 0.025; Test type: Superiority or Other; p < 0.001, ANCOVA — Hypotheses were tested in a sequential fashion using a gatekeeping strategy and adjusted for multiplicity. Statistical significance at 0.05 level was required for this variable; Change from baseline ANCOVA model: treatment group, baseline value, pooled site. Baseline-by-treatment interaction included if interaction at p<0.10

2. Primary Outcome: Improvement in the Sexual Quality of Life in the Subject and His Study Partner as Measured by the Sexual Quality of Life (SQoL) Domain of the Sexual Life Quality Questionnaire (SLQQ)
Description: The original item scores (-4 to 4 range) were converted to 0 to 8 scale score by adding 4 to each recorded responses. Each transformed score was multiplied by 12.5 for a total range of 0 to 100. Higher scores are indicative of a higher sexual quality of life.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 72 | 244
units on a scale
  SQoL - Subject (change from baseline) | 12.59 (2.866) | 39.37 (1.651)
  SQoL-Partner (change from baseline) (n=70, n=238) | 7.93 (2.861) | 32.87 (1.638)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Subject. Hypotheses were tested in a sequential fashion using a gatekeeping strategy and adjusted for multiplicity. To adjust for multiplicity, statistical significance at 0.025 level was required for this variable; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Tadalafil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Partner. Hypotheses were tested in a sequential fashion using a gatekeeping strategy and adjusted for multiplicity. To adjust for multiplicity, statistical significance at 0.025 level was required for this variable; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline to Week 12 Endpoint in the International Index of Erectile Function - Intercourse Satisfaction Domain - Subject Response
Description: Self-reported intercourse satisfaction over the past 4 weeks. Scores range from 0 (low/no satisfaction to 5 (high satisfaction), thus the 3 questions of the IIEF-IS domain range from 0 to 15.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 72 | 244
units on a scale | 0.09 (0.356) | 2.74 (0.205)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Overall Satisfaction Domain of the International Index of Erectile Function (IIEF-OS) - Subject Response
Description: Self-reported overall satisfaction over the past 4 weeks. Scores range from 0 (low/no satisfaction to 5 (high satisfaction), thus the 2 questions of the IIEF-OS domain range from 0 to 10.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 72 | 244
units on a scale | 0.44 (0.257) | 2.57 (0.148)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Sexual Life Quality Questionnaire (SLQQ) Treatment Satisfaction Domain
Description: The 6 SLQQ-treatment satisfaction questions were answered by subject and partner at Visit 4/Final Visit. Original item scores (1 to 6 range) were converted to 0 to 5 scale by subtracting 1 to each recorded responses. Each transformed score was multiplied by 20. Total range of scores: 0 (low satisfaction) to 100 (high satisfaction).
Time Frame: 12 weeks
Population: all randomized participants having post-baseline data measurement on this variable
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 72 | 244
units on a scale
  SLQQ - Subject (n=72, n=244) | 51.58 (2.246) | 75.04 (1.293)
  SLQQ - Partner (n=70, n=238) | 55.25 (2.115) | 73.42 (1.214)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value is for subject scores; ANCOVA included:treatment, baseline value of IIEF EF Domain, pooled site. Baseline-value-by-treatment interaction included if interaction at p<0.10
Statistical Analysis 2: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value is for partner scores; [statistical method as in outcome 5, analysis 1]

6. Primary Outcome: Change From Baseline to Endpoint in the Percent of "Yes" Responses to Sexual Encounter Profile (SEP) Diary Questions 2 (SEP2) and 3 (SEP3).
Description: The baseline and endpoint score for each SEP question 2 (Insert penis into vagina) and 3 (Successful intercourse) are the subject's percentage of "yes" responses to those questions during the run-in period and postbaseline period, respectively.
Time Frame: Baseline and 12 weeks
Population: all randomized participants having both baseline and at least one post-baseline data measurement
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 74 | 251
percent
  Question 2 change from baseline in percent "yes" | 2.19 (2.833) | 28.80 (1.644)
  Question 3 change from baseline in percent "yes" | 10.80 (3.767) | 46.46 (2.185)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for SEP Question 2. Hypotheses were tested in a sequential fashion using a gatekeeping strategy and adjusted for multiplicity. Statistical significance at 0.05 level was required for this variable; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Tadalafil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for SEP Question 3. Hypotheses were tested in a sequential fashion using a gatekeeping strategy and adjusted for multiplicity. Statistical significance at 0.05 level was required for this variable; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Percent of "Yes" Responses to Sexual Encounter Profile (SEP) Questions 4 and 5 - Subject Response
Description: The baseline and endpoint score for each SEP question 4 (Satisfied with hardness) and 5 (Satisfied overall) are the subject's percentage of "yes" responses to those questions during the run-in period and postbaseline period, respectively.
Time Frame: Baseline and 12 weeks
Population: all randomized participants having both baseline and at least one post-baseline data measurement
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 74 | 251
percent
  Question 4 change from baseline in percent "Yes" | 12.08 (3.936) | 50.05 (2.283)
  Question 5 change from baseline in percent "Yes" | 11.47 (3.951) | 48.78 (2.292)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value for SEP Question 4; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value for SEP Question 5; [statistical method as in outcome 1, analysis 1]

8. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Percent of "Yes" Responses to Partner-Sexual Encounter Profile (SEP) Question 3 - Partner Response
Description: The baseline and endpoint score for partner SEP question 3 (Satisfied overall) are the partner's percentage of "yes" responses to the question during the run-in period and postbaseline period, respectively.
Time Frame: Baseline and 12 weeks
Population: all randomized participants having both baseline and at least one post-baseline data measurement
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 73 | 250
percent | 10.21 (3.595) | 43.16 (2.072)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]

9. Secondary Outcome: Change From Baseline to 12 Week Endpoint in the Satisfaction Domain of the Female Sexual Function Index (FSFI) - Partner Response
Description: The FSFI Satisfaction Domain (items 14-16) measures satisfaction with emotional closeness, sexual relationship, and overall sexual life. Each question is scored on a 0/1 to 5 scale and domain score is calculated by multiplying the total points by 0.4, for a total score range of 0.8 to 6, with higher scores indicating greater satisfaction.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 70 | 238
units on a scale | -0.40 (0.130) | 0.32 (0.075)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]

10. Secondary Outcome: Percent of Subjects With "Yes" Responses to Global Assessment Questionnaire (GAQ) - Subject Response
Description: Percent of subjects with "Yes" responses to Question 1 (Improvement in Erections) and Question 2 (Improvement in the Ability to Engage in Sexual Activity)
Time Frame: 12 weeks
Population: all randomized participants having post-baseline data measurement on this variable
Measure: Number; unit: percentage of subjects answering Yes
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 72 | 244
percentage of subjects answering Yes
  GAQ Question 1 | 26 | 81
  GAQ Question 2 | 22 | 79
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value is for GAQ Question 1; Model included:treatment, baseline value of IIEF EF Domain, pooled site. Baseline-value-by-treatment interaction included if interaction at p<0.10
Statistical Analysis 2: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value is for GAQ Question 2; [statistical method as in outcome 10, analysis 1]

11. Secondary Outcome: Percent of Partners With "Yes" Responses to Global Assessment Questionnaire (GAQ) - Partner Response
Description: Percent of Partners with "Yes" responses to Question 1 (Improvement in Erections) and Question 2 (Improvement in the Ability to Engage in Sexual Activity)
Time Frame: 12 weeks
Population: all randomized participants having post-baseline data measurement on this variable
Measure: Number; unit: percentage of partners answering Yes
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 70 | 238
percentage of partners answering Yes
  GAQ Question 1 | 30 | 79
  GAQ Question 2 | 24 | 76
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value is for GAQ Question 1; [statistical method as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value is for GAQ Question 2; [statistical method as in outcome 10, analysis 1]

12. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Percent of "Yes" Responses to Partner-Sexual Encounter Profile (SEP) Questions 1 and 2 - Partner Response
Description: The baseline and endpoint score for each SEP question 1 (Achieve some erection) and 2 (Insert penis into vagina) are the partner's percentage of "yes" responses to those questions during the run-in period and postbaseline period, respectively.
Time Frame: Baseline and 12 weeks
Population: all randomized participants having both baseline and at least one post-baseline data measurement
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 73 | 250
percent
  Question 1 change from baseline in percent "Yes" | 1.25 (2.224) | 18.34 (1.270)
  Question 2 change from baseline in percent "Yes" | 6.97 (2.896) | 30.69 (1.662)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for SEP Question 1; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for SEP Question 2; [statistical method as in outcome 1, analysis 1]

13. Secondary Outcome: Change From Baseline to 12 Week Endpoint in the Self-Esteem and Relationship (SEAR) Questionnaire
Description: Measures improvement in self-esteem and relationship satisfaction. Questionnaire consists of two domains, Sexual Relationship (items 1-8) and Confidence (items 9-14). Overall score is transformed onto a 0 (least favorable) to 100 (most favorable) scale. Overall score was calculated from two domains and subscales scores.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 72 | 244
units on a scale
  Total Score change from baseline | 3.07 (2.616) | 30.44 (1.506)
  Sexual Relationship change from baseline | 4.61 (2.903) | 34.28 (1.673)
  Confidence change from baseline | 0.91 (2.567) | 25.35 (1.475)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for SEAR Total Score; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for SEAR Sexual Relationship; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for SEAR Confidence; [statistical method as in outcome 1, analysis 1]

14. Secondary Outcome: Change From Baseline to 12 Week Endpoint in the Self-Esteem and Relationship (SEAR) Questionnaire - Confidence Domain Subscales
Description: Measures improvement in confidence (items 9-14). Confidence domain consists of two subscales (Self-Esteem, items 9-12; Overall Relationship, items 13 and 14). Each domain score, subscale score, and overall score are transformed onto a 0 (least favorable) to 100 (most favorable) scale.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 72 | 244
units on a scale
  Self-Esteem change from baseline | 3.26 (2.743) | 29.56 (1.579)
  Overall Relationship change from baseline | -4.04 (2.792) | 16.97 (1.603)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for SEAR Self-Esteem; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for SEAR Overall Relationship; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Placebo | Tadalafil
Serious Adverse Events (participants affected / at risk) | 1 | 3
Other Adverse Events (participants affected / at risk) | 21 | 77
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | Tadalafil
Pancreatitis (Gastrointestinal disorders) | 1/78 (1) | 0/264 (0)
Hypersensitivity (Immune system disorders) | 0/78 (0) | 1/264 (1)
Gastroenteritis (Infections and infestations) | 0/78 (0) | 1/264 (1)
Cerebrovascular accident (Nervous system disorders) | 0/78 (0) | 1/264 (1)
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | Tadalafil
Hypoacusis (Ear and labyrinth disorders) | 0/78 (0) | 1/264 (1)
Hypogonadism (Endocrine disorders) | 0/78 (0) | 1/264 (1)
Blepharitis (Eye disorders) | 0/78 (0) | 1/264 (1)
Conjunctivitis (Eye disorders) | 0/78 (0) | 1/264 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0/78 (0) | 1/264 (1)
Constipation (Gastrointestinal disorders) | 1/78 (1) | 0/264 (0)
Diarrhoea (Gastrointestinal disorders) | 1/78 (1) | 5/264 (5)
Dry mouth (Gastrointestinal disorders) | 1/78 (1) | 0/264 (0)
Dyspepsia (Gastrointestinal disorders) | 0/78 (0) | 12/264 (13)
Dysphagia (Gastrointestinal disorders) | 0/78 (0) | 1/264 (1)
Gastritis (Gastrointestinal disorders) | 0/78 (0) | 2/264 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0/78 (0) | 5/264 (5)
Hiatus hernia (Gastrointestinal disorders) | 0/78 (0) | 1/264 (1)
Nausea (Gastrointestinal disorders) | 0/78 (0) | 3/264 (3)
Toothache (Gastrointestinal disorders) | 0/78 (0) | 1/264 (1)
Vomiting (Gastrointestinal disorders) | 1/78 (1) | 2/264 (2)
Chest pain (General disorders) | 0/78 (0) | 1/264 (1)
Discomfort (General disorders) | 0/78 (0) | 1/264 (1)
Fatigue (General disorders) | 2/78 (2) | 0/264 (0)
Oedema mucosal (General disorders) | 0/78 (0) | 1/264 (1)
Pyrexia (General disorders) | 0/78 (0) | 1/264 (1)
Drug hypersensitivity (Immune system disorders) | 1/78 (1) | 0/264 (0)
Amoebic dysentery (Infections and infestations) | 0/78 (0) | 1/264 (1)
Anogenital warts (Infections and infestations) | 0/78 (0) | 1/264 (1)
Bronchitis (Infections and infestations) | 1/78 (1) | 0/264 (0)
Gastroenteritis (Infections and infestations) | 3/78 (3) | 2/264 (3)
Herpes simplex (Infections and infestations) | 1/78 (1) | 0/264 (0)
Herpes zoster (Infections and infestations) | 0/78 (0) | 1/264 (1)
Influenza (Infections and infestations) | 0/78 (0) | 2/264 (2)
Nasopharyngitis (Infections and infestations) | 0/78 (0) | 2/264 (2)
Onychomycosis (Infections and infestations) | 0/78 (0) | 1/264 (1)
Oral herpes (Infections and infestations) | 0/78 (0) | 1/264 (1)
Pharyngitis (Infections and infestations) | 1/78 (1) | 3/264 (4)
Rhinitis (Infections and infestations) | 0/78 (0) | 3/264 (3)
Sinusitis (Infections and infestations) | 1/78 (1) | 0/264 (0)
Tonsillitis (Infections and infestations) | 1/78 (1) | 3/264 (3)
Tooth infection (Infections and infestations) | 1/78 (1) | 0/264 (0)
Wound (Injury, poisoning and procedural complications) | 0/78 (0) | 1/264 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1/78 (1) | 0/264 (0)
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 1/78 (1) | 0/264 (0)
Gout (Metabolism and nutrition disorders) | 0/78 (0) | 1/264 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1/78 (1) | 0/264 (0)
Obesity (Metabolism and nutrition disorders) | 0/78 (0) | 1/264 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/78 (0) | 1/264 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1/78 (2) | 5/264 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1/78 (1) | 3/264 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1/78 (1) | 0/264 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0/78 (0) | 4/264 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/78 (0) | 1/264 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0/78 (0) | 5/264 (5)
Dizziness (Nervous system disorders) | 1/78 (1) | 1/264 (1)
Headache (Nervous system disorders) | 3/78 (4) | 22/264 (26)
Hypoaesthesia (Nervous system disorders) | 0/78 (0) | 1/264 (1)
Sciatica (Nervous system disorders) | 0/78 (0) | 1/264 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/78 (0) | 1/264 (1)
Anxiety (Psychiatric disorders) | 0/78 (0) | 1/264 (1)
Insomnia (Psychiatric disorders) | 1/78 (1) | 0/264 (0)
Libido decreased (Psychiatric disorders) | 0/78 (0) | 1/264 (1)
Pollakiuria (Renal and urinary disorders) | 0/78 (0) | 1/264 (1)
Ejaculation delayed (Reproductive system and breast disorders) | 0/78 (0) | 1/264 (1)
Gynaecomastia (Reproductive system and breast disorders) | 0/78 (0) | 1/264 (1)
Hypoaesthesia of genital male (Reproductive system and breast disorders) | 0/78 (0) | 1/264 (1)
Painful erection (Reproductive system and breast disorders) | 0/78 (0) | 1/264 (2)
Testicular pain (Reproductive system and breast disorders) | 1/78 (1) | 0/264 (0)
Varicocele (Reproductive system and breast disorders) | 0/78 (0) | 1/264 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1/78 (1) | 1/264 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/78 (0) | 1/264 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0/78 (0) | 1/264 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0/78 (0) | 7/264 (9)
Erythema (Skin and subcutaneous tissue disorders) | 1/78 (1) | 1/264 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1/78 (1) | 0/264 (0)
Rash (Skin and subcutaneous tissue disorders) | 0/78 (0) | 1/264 (1)
Dental prosthesis placement (Surgical and medical procedures) | 0/78 (0) | 1/264 (1)
Hot flush (Vascular disorders) | 0/78 (0) | 2/264 (2)
Hypertension (Vascular disorders) | 0/78 (0) | 3/264 (3)
Hypotension (Vascular disorders) | 1/78 (1) | 0/264 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days